CLINICAL TRIAL: NCT06325111
Title: Exploring Genetic, Epigenetic and Environmental Determinants of Glycaemic Control in Children and Young Individuals With Type 1 Diabetes
Brief Title: Determinants of Glycaemic Control in Children With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 06/2023
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes glycaemic control; Epigenetic modifications; Diabetes-related complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with T1D and optimal glycaemic control: Optimal glycaemic control will be defined as HbA1c values <7%
  Interventions: Other: Determinants of T1D glycaemic control
- Patients with T1D and poor glycaemic control: Poor glycemic control will be defined as HbA1c value ≥7%
  Interventions: Other: Determinants of T1D glycaemic control

INTERVENTIONS:
Other: Determinants of T1D glycaemic control — DNA genotyping, microbiome, DNA methylation and microRNAs analysis

SUMMARY:
Type 1 diabetes (T1D) is a common chronic disease of childhood associated with a significantly increased risk of micro- and macro-vascular complications, including neuropathy, nephropathy and cardiovascular diseases. The risk of development T1D comorbidities is associated with glycaemic control, a complex mechanism involving biological, physiological environmental factors.

While more than 60 genetic variants were already associated with Glycated hemoglobin (HbA1c) in healthy subjects, very few genes have been identified in T1D individuals. Also, hyperglycaemia could be the cause of epigenetic changes at specific target genes, such as DNA methylation, histone modifications and microRNAs, correlated to accelerated development of diabetes-related complications. Most recently, increasing evidence also suggested that human microbiome may play a crucial role in the onset and progression of T1D and dysbiosis of the gut and oral microbiota was reported as a typical feature of hyperglycaemia.

However, potential differences among poorly and good managed T1D subjects have not been still studied. Also, the exact mechanism by long-term hyperglycaemia's acts in T1D remains poorly understood. Therefore, this project will explore an emerging area of research by the study of possible genetic, epigenetic and environmental biomarkers among T1D subjects with different glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes subjects
* Age from 6 to 20 years old
* At least 5 years of duration of disease

Exclusion Criteria:

* Type 1 diabetes subjects incapable of giving valid informed consent or whose parents are incapable of giving valid informed consent.
* Type 1 diabetes subjects for whom it is not possible to collect information on the clinical history, starting from the onset of diabetes
* Subjects with other types of diabetes (i.e. type 2, monogenic diabetes, cystic fibrosis related diabetes)

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: T1D subjects (children and young adults) attending to several Diabetes Units of Italian and European institutions
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Identification of genes involved in T1D glycaemic control | Through study completion, an average of 18 months
  DNA will be isolated from saliva by Genefix Saliva DNA/RNA collection kit (Isohelix, UK) and whole genome genotyping will be performed using Illumina chip arrays (CA, USA).
Identification of DNA methylation patterns involved in T1D glycaemic control | Through study completion, an average of 18 months
  Peripheral blood will be collected from each participant into EDTA-containing tubes and Genome-wide DNA methylation will be performed using the Illumina Infinium Human Methylation EPIC BeadChip array
Identification of microRNAs involved in T1D glycaemic control | Through study completion, an average of 18 months
  Peripheral blood will be collected from each participant into Ethylenediaminetetraacetic acid (EDTA)-containing tubes for microRNAs sequencing. Illumina TruSeq Small RNA Sample Preparation kit will be used for library preparation, and sequencing will be conducted by Illumina platform (CA, USA).
Identification of oral microbiome characteristics associated to T1D glycaemic control | Through study completion, an average of 18 months
  Bacterial DNA will be extracted from saliva and a 500 base pair region of the V1-V3 portion of the 16S ribosomal RNA gene as well as the 200 base pair region of the V3 portion will be amplified. The V3 amplicon will be used for template preparation and will be sequenced using the Ion PGM Hi-Q View sequencing kit (Life Technologies, New York, NY, USA) with the IonPGM™System technology

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided